CLINICAL TRIAL: NCT03525119
Title: A Randomized, Observer Blind, Phase 3 Trial to Investigate the Immunogenicity and Safety of the Co-administration of a Subcutaneous Tetravalent Dengue Vaccine Candidate (TDV) and an Intramuscular Hepatitis A Virus (Inactivated) Vaccine in Healthy Subjects Aged 18 to 60 Years in Non-endemic Country(Ies) for Dengue
Brief Title: Immunogenicity and Safety of Tetravalent Dengue Vaccine (TDV) Co-administered With an Hepatitis A Virus Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DEN-314; 2017-001071-23 (EudraCT Number); U1111-1192-7761 (Other: WHO); 18/NW/0008 (Registry Identifier: NRES)
Record Dates: First submitted 2018-04-27; First posted 2018-05-15 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Healthy Volunteers
Keywords: Vaccine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HAV Vaccine 1.0 ml + Placebo/ Placebo (Other): HAV vaccine 1.0 ml, injection, IM, and placebo-matching injection, SC, once on Day 1 (first dose) followed by placebo-matching injection, SC on Day 90 (second dose).
  Interventions: Biological: HAV Vaccine; Biological: TDV Placebo
- TDV 0.5 ml + Placebo/ TDV 0.5 ml (Experimental): TDV 0.5 ml, injection, SC, and placebo-matching injection, IM, once on Day 1 (first dose) followed by TDV 0.5 ml, injection, SC on Day 90 (second dose).
  Interventions: Biological: TDV; Biological: HAV Vaccine Placebo
- TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml (Experimental): TDV 0.5 ml, injection, SC, and HAV vaccine 1.0 ml, injection, IM, once on Day 1 (first dose) followed by TDV 0.5 ml, injection, SC on Day 90 (second dose).
  Interventions: Biological: TDV; Biological: HAV Vaccine

INTERVENTIONS:
Biological: TDV — TDV SC injection
  Arms: TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml; TDV 0.5 ml + Placebo/ TDV 0.5 ml
Biological: HAV Vaccine — HAV Vaccine IM injection.
  Arms: HAV Vaccine 1.0 ml + Placebo/ Placebo; TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Biological: TDV Placebo — Placebo-matching (normal saline (0.9% NaCl) SC injection.
  Arms: HAV Vaccine 1.0 ml + Placebo/ Placebo
Biological: HAV Vaccine Placebo — Placebo-matching (normal saline (0.9% NaCl) IM injection.
  Arms: TDV 0.5 ml + Placebo/ TDV 0.5 ml

SUMMARY:
The purpose of this study is to investigate the immunogenicity and safety of the concomitant administration of TDV (subcutaneous [SC] injection) and of hepatitis A virus (HAV) vaccine (intramuscular [IM] injection) in healthy participants aged 18 to 60 years living in country(ies) non-endemic for both dengue and hepatitis.

DETAILED DESCRIPTION:
The vaccine tested in this study is TDV. TDV co-administered with HAV vaccine will be tested to assess immunogenicity and safety in healthy participants in non-endemic area(s) for dengue and HAV.

The study will enroll approximately 900 patients. Participants will be randomly assigned to one of the three groups-which will remain undisclosed to the observer. Participants will be randomized in 1:1:1 ratio to receive:

* Group 1: HAV vaccine (IM) and TDV placebo-matching injection (SC), co-administered at Day 1 (Month 0 [M0]); TDV placebo-matching injection (SC) administered at Day 90 (Month 3 [M3])
* Group 2: TDV (SC) and HAV placebo-matching injection (IM), co-administered at Day 1 (Month 0 [M0]); TDV (SC) administered at Day 90(Month 3 [M3])
* Group 3: TDV (SC) and HAV vaccine (IM), co-administered at Day 1 (Month 0 [M0]); TDV (SC) administered at Day 90 (Month 3 [M3])

This multi-center trial will be conducted in United Kingdom. The overall time to participate in this study is 270 days. Participants will have multiple visits to the clinic with a 6-months follow up after the last study administration, including a final visit at Day 270.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is aged 18 to 60 years, inclusive.
2. Participants who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and the clinical judgment of the Investigator.
3. The participant signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
4. Participants who can comply with trial procedures and are available for the duration of follow-up.

Exclusion Criteria:

1. Participants with an elevated oral temperature (≥38°C or 100.4°F) within 3 days of the intended date of vaccination.
2. Known hypersensitivity or allergy to any of the vaccine components (including excipients of the investigational vaccines or placebo).
3. Participants with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the participant's ability to participate in the trial.
4. Participants with any history of progressive or severe neurologic disorder, seizure disorder orneuro-inflammatory disease (eg, Guillain-Barré syndrome).
5. Participants with history or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose additional risk to the participant due to participation in the trial.
6. Known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥ 2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (Month 0).
   3. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (Month 0) or planned administration during the trial.
   4. Receipt of immunostimulants within 60 days prior to Day 1 (Month 0).
   5. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (Month 0).
   6. Human immunodeficiency virus (HIV) infection or HIV-related disease.
   7. Hepatitis A virus (HAV) infection.
   8. Hepatitis C virus infection.
   9. Genetic immunodeficiency.
7. Abnormalities of splenic or thymic function.
8. Participants with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
9. Participants with any serious chronic or progressive disease according to judgment of the Investigator (eg, neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
10. Participants with body mass index (BMI) greater than or equal to 35 kg/m^2 (=weight in kg/[height in meters^2]).
11. Participants participating in any clinical trial with another investigational product 30 days prior to Day 1 (Month 0) or intent to participate in another clinical trial at any time during the conduct of this trial.
12. Participants who received any other vaccine within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of trial vaccine administration.
13. Previous HAV vaccination (in a clinical trial or with an approved product).
14. Participants involved in the trial conduct or their first degree relatives.
15. Participants with history of substance or alcohol abuse within the past 2 years.
16. Female participants who are pregnant or breastfeeding.
17. Females of childbearing potential who are sexually active, and who have not used any of the acceptable contraceptive methods for at least 2 months prior to Day 1 (Month 0).

    1. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: bilateral tubal ligation (at least 1 year previously), bilateral oophorectomy (at least 1 year previously) or hysterectomy
    2. Acceptable birth control methods are defined as one or more of the following:

    i. Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring).

    ii. Barrier method (condom with spermicide or diaphragm with spermicide) each and every time during intercourse.

    iii. Intrauterine device (IUD). iv. Monogamous relationship with vasectomized partner (partner must have been vasectomized for at least 6 months prior to Day 1 [Month 0]).

    Other contraceptive methods may be considered in agreement with the Sponsor and implemented only after approval of a substantial amendment by the regulatory authorities and by the appropriate ethics committee.
18. Females of childbearing potential who are sexually active, and who refuse to use an acceptable contraceptive method up to 6 weeks after the last dose of trial vaccine (Day 90 [M3]). In addition, they must be advised not to donate ova during this period.
19. Any positive or indeterminate pregnancy test.
20. Previous and planned vaccination (during the trial conduct) against any flaviviruses including dengue, yellow fever (YF), Japanese Encephalitis (JE) viruses or tick-borne encephalitis.
21. Previous participation in any clinical trial of a dengue or other flavivirus (eg, West Nile [WN] virus) candidate vaccine, except for participants who received placebo in those trials.
22. Participants with a current or previous infection with a flavivirus such as dengue, Zika, YF, JE, WN fever, tick-borne encephalitis or Murray Valley encephalitis and participants with a history of prolonged (≥1 year) habitation in a dengue endemic area.
23. Participants with contraindications, warnings and/or precautions to vaccination with the HAV vaccine as specified within the product information.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (10):
- United Kingdom (10):
  - Synexus - Midlands, Edgbaston, Birmingham
  - Synexus - Lancashire, Chorley, Lancashire
  - Synexus - Merseyside, Waterloo, Liverpool
  - Royal Hallamshire Hospital, Sheffield, Yorkshire
  - Synexus - Wales, Cardiff
  - Synexus - Scotland, Glasgow
  - North East Clinical Research Centre, Hexham General Hospital, Hexham
  - Synexus - Manchester, Manchester
  - Synexus - Thames Valley, Reading
  - North Tees Clinical Research Centre, Middlefield Centre, University Hospital of North Tees, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.

REFERENCES:
- [Derived] Tricou V, Eyre S, Ramjee M, Collini P, Mojares Z, Loeliger E, Mandaric S, Rauscher M, Brose M, Lefevre I, Folschweiller N, Wallace D. A randomized phase 3 trial of the immunogenicity and safety of coadministration of a live-attenuated tetravalent dengue vaccine (TAK-003) and an inactivated hepatitis a (HAV) virus vaccine in a dengue non-endemic country. Vaccine. 2023 Feb 10;41(7):1398-1407. doi: 10.1016/j.vaccine.2023.01.007. Epub 2023 Jan 19. PMID 36681529
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b60224db2bf003ab4969e?idFilter=%5B%22DEN-314%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in United Kingdom from 16-May-2018 to 09-Jul-2019.
Pre-assignment Details: Healthy participants were randomized in 1:1:1 ratio in 3 parallel groups: Group 1 received 1 dose of Hepatitis A Virus (HAV) vaccine and Tetravalent Dengue Vaccine Candidate (TDV) placebo matching injection, Group 2 received 2 doses of TDV and HAV vaccine placebo matching injection and Group 3 received 1 dose of HAV vaccine and 2 doses of TDV.
Period: Overall Study
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Started | 300 | 300 | 300
Safety Population (Received at Least 1 Vaccination with Investigational Products (IPs) i.e. HAV vaccine/placebo/TDV) | 299 | 300 | 298
Completed | 260 | 261 | 257
Not Completed | 40 | 39 | 43
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 32 | 33 | 37
Not completed — Withdrawal by Subject | 5 | 4 | 2
Not completed — Reason not Specified | 2 | 1 | 2
Not completed — Randomized but not Vaccinated | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants enrolled and randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml | Total
Number analyzed (Participants) | 300 | 300 | 300 | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (12.03) | 36.0 (11.88) | 35.5 (11.94) | 35.4 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 120 | 90 | 317
  Male | 193 | 180 | 210 | 583
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 1 | 11
  Not Hispanic or Latino | 290 | 293 | 296 | 879
  Unknown or Not Reported | 4 | 3 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 5 | 9 | 11 | 25
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 6 | 4 | 6 | 16
  White | 280 | 281 | 279 | 840
  More than one race | 7 | 4 | 4 | 15
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 300 | 300 | 300 | 900
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available at Baseline.
  cm
    number analyzed (Participants) | 299 | 300 | 297 | 896
    (all) | 173.80 (9.299) | 172.12 (9.163) | 173.00 (9.110) | 172.97 (9.207)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with data available at Baseline.
  kg
    number analyzed (Participants) | 299 | 300 | 297 | 896
    (all) | 79.24 (15.547) | 78.18 (15.570) | 78.92 (15.243) | 78.78 (15.444)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight/Height. Population: Number analyzed is the number of participants with data available at Baseline.
  kg/m^2
    number analyzed (Participants) | 299 | 300 | 297 | 896
    (all) | 26.16 (4.256) | 26.31 (4.354) | 26.29 (4.283) | 26.25 (4.293)
Baseline Seroprotection Against HAV [Count of Participants; unit: Participants] — Seroprotection was defined as serum anti-HAV antibody levels ≥12.5 mIU/mL, measured by Enzyme-Linked Immunosorbent Assay (ELISA). Population: Number analyzed is the number of participants from Immunogenicity Subset, with data available for analyses at Baseline.
  Participants
    number analyzed (Participants) | 118 | 121 | 122 | 361
    Yes | 31 | 38 | 30 | 99
    No | 87 | 83 | 92 | 262
Baseline Seropositivity Status for Dengue [Count of Participants; unit: Participants] — Seropositivity defined as a reciprocal neutralizing titer >=10 for at least 1 dengue serotype. Seronegativity was defined as having a reciprocal neutralizing titer <10 for all dengue serotypes. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4. Population: Number analyzed is the number of participants from Immunogenicity Subset, with data available for analyses at Baseline.
  Participants
    number analyzed (Participants) | 118 | 119 | 120 | 357
    Seropositive | 11 | 8 | 9 | 28
    Seronegative | 107 | 111 | 111 | 329
Baseline Seropositivity Rate for Each Dengue Serotype [Count of Participants; unit: Participants] — Seropositivity rate, defined as the percentage of participants seropositive for the given dengue serotype, derived from the titers of dengue-neutralizing antibodies. Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4. Population: Number analyzed is the number of participants from Immunogenicity Subset, with data available for analyses at Baseline. Participants are repeated across categories as seropositivity for more than serotype is reported.
  Participants
    DENV-1: number analyzed (Participants) | 118 | 119 | 120 | 357
    DENV-1 | 6 | 6 | 5 | 17
    DENV-2: number analyzed (Participants) | 118 | 119 | 120 | 357
    DENV-2 | 4 | 2 | 5 | 11
    DENV-3: number analyzed (Participants) | 118 | 119 | 120 | 357
    DENV-3 | 4 | 1 | 1 | 6
    DENV-4: number analyzed (Participants) | 118 | 119 | 120 | 357
    DENV-4 | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants HAV/Dengue Virus (DENV)-Naive at Baseline Who Are Seroprotected Against HAV at Day 30
Description: Seroprotection is defined as serum anti-HAV antibody levels ≥12.5 mIU/mL, measured by enzyme-linked immunosorbent assay (ELISA). Immunological naivety to HAV/DENV is defined as anti-HAV antibody levels <12.5 mIU/mL and reciprocal neutralizing titers for all 4 dengue serotypes <10. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: One month post first vaccination (Day 30)
Population: HAV PPS: All HAV & DENV-naïve participants in the immunogenicity subset who received at least 1 dose of trial vaccine, with available Day 1 and Day 30 HAV immunogenicity measurements, and who have no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 68 | 66 | 79
percentage of participants | 97.1 [89.8 to 99.6] | 9.1 [3.4 to 18.7] | 98.7 [93.1 to 100.0]
Statistical Analysis 1: Comparison: HAV Vaccine 1.0 ml + Placebo/ Placebo vs TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml; Test type: Non-Inferiority — As per predefined criteria in protocol the non-inferiority was established only between group 1 and group 3. Non-inferiority of HAV+TDV to HAV was established if the upper bound of the 95% CI was less than 10%; Seroprotection Rate Difference = -1.68, 95% CI 2-sided [-8.91 to 4.28]

2. Secondary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Day 30 and Day 120 in Participants HAV/DENV-naive at Baseline
Description: GMTs of neutralizing antibodies were measured by microneutralization test 50% [MNT50] for each of the 4 Dengue Serotypes. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: One month post first vaccination (Day 30) and one month post second vaccination (Day 120)
Population: TDV PPS: All HAV & DENV-naïve participants in the immunogenicity subset who received at least 1 dose of trial vaccine, with available Day 1 and at least 1 post-dose immunogenicity measurements, and who have no major protocol violations. Number analyzed are participants with data available at the given timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 66 | 63 | 67
titer
  DENV 1, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 1, Day 30 | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the lower limit of detection (LLOD). | 108.2 [69.2 to 169.1] | 152.5 [104.4 to 222.8]
  DENV 2, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 2, Day 30 | 6.0 [5.1 to 7.1] | 2897.9 [1469.2 to 5715.6] | 3960.0 [2310.7 to 6786.5]
  DENV 3, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 3, Day 30 | 5.3 [4.7 to 5.8] | 95.4 [59.5 to 153.2] | 140.5 [96.8 to 203.9]
  DENV 4, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 4, Day 30 | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 74.3 [49.0 to 112.9] | 142.1 [90.5 to 223.2]
  DENV 1, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 1, Day 120 | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 171.3 [104.5 to 281.0] | 173.7 [120.1 to 251.3]
  DENV 2, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 2, Day 120 | 5.7 [4.9 to 6.7] | 2064.1 [1459.7 to 2918.9] | 1764.3 [1238.6 to 2513.0]
  DENV 3, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 3, Day 120 | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 83.8 [59.0 to 119.0] | 92.6 [71.3 to 120.3]
  DENV 4, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 4, Day 120 | 5.0 [NA to NA] — Lower and upper limits of CI could not be evaluated as titers were below the LLOD. | 56.1 [41.0 to 76.7] | 81.4 [59.2 to 111.8]

3. Secondary Outcome: Percentage of Participants HAV/DENV-naive at Baseline Who Are Seropositive for Each of the 4 Dengue Serotypes at Day 30 and Day 120
Description: Seropositivity is defined as a reciprocal neutralizing titer ≥10. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: One month post first vaccination (Day 30) and one month post second vaccination (Day 120)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 66 | 63 | 67
percentage of participants
  DENV 1, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 1, Day 30 | 0 [0.0 to 5.9] | 88.3 [77.4 to 95.2] | 95.4 [87.1 to 99.0]
  DENV 2, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 2, Day 30 | 8.2 [2.7 to 18.1] | 91.7 [81.6 to 97.2] | 96.9 [89.3 to 99.6]
  DENV 3, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 3, Day 30 | 1.6 [0.0 to 8.8] | 85.0 [73.4 to 92.9] | 95.4 [87.1 to 99.0]
  DENV 4, Day 30: number analyzed (Participants) | 61 | 60 | 65
  DENV 4, Day 30 | 0 [0.0 to 5.9] | 86.7 [75.4 to 94.1] | 90.8 [81.0 to 96.5]
  DENV 1, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 1, Day 120 | 0 [0.0 to 7.1] | 100.0 [93.5 to 100.0] | 100.0 [94.2 to 100.0]
  DENV 2, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 2, Day 120 | 6.0 [1.3 to 16.5] | 100.0 [93.5 to 100.0] | 100.0 [94.2 to 100.0]
  DENV 3, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 3, Day 120 | 0 [0.0 to 7.1] | 92.7 [82.4 to 98.0] | 98.4 [91.3 to 100.0]
  DENV 4, Day 120: number analyzed (Participants) | 50 | 55 | 62
  DENV 4, Day 120 | 0 [0.0 to 7.1] | 96.4 [87.5 to 99.6] | 96.8 [88.8 to 99.6]

4. Secondary Outcome: Geometric Mean Concentrations (GMC) of Anti-HAV Antibodies at Day 30 in Participants HAV/DENV-naive at Baseline
Description: GMC of anti-HAV antibodies were measured by ELISA.
Time Frame: One month post first vaccination (Day 30)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 68 | 66 | 79
mIU/mL | 82.1 [62.9 to 107.1] | 6.7 [6.4 to 7.2] | 93.0 [76.1 to 113.6]

5. Secondary Outcome: Percentage of Participants With Solicited (Local Injection) Site Adverse Events (AEs) by Severity After Each Vaccination
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain (none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents daily activity with or without treatment), redness (erythema) (<2.5 cm, mild: 2.5-5 cm, moderate: >5 to <=10 cm, severe: >10 cm) and swelling (edema/induration) (<2.5 cm, mild: 2.5-5 cm, moderate: >5 to <=10 cm, severe: >10 cm ). The percentages were rounded off to the first decimal place.
Time Frame: Within 7 days after each vaccination
Population: Safety Set included all participants who received at least 1 dose of trial vaccine. Number analyzed is the number of participants with data available for the specific category. Only categories for which there was at least 1 participant are reported.
Measure: Number; unit: percentage of participants
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 299 | 300 | 298
percentage of participants
  After First Vaccination IM,Any Local AEs: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination IM,Any Local AEs | 45.0 | 15.4 | 49.1
  After First Vaccination, IM, Pain-Any: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, IM, Pain-Any | 44.6 | 14.4 | 48.4
  After First Vaccination, IM, Pain-Mild: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, IM, Pain-Mild | 38.1 | 13.0 | 43.9
  After First Vaccination, IM, Pain-Moderate: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, IM, Pain-Moderate | 6.6 | 1.0 | 4.2
  After First Vaccination, IM, Pain-Severe: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, IM, Pain-Severe | 0 | 0.3 | 0.4
  After First Vaccination, IM, Erythema-Any: number analyzed (Participants) | 287 | 291 | 285
  After First Vaccination, IM, Erythema-Any | 2.4 | 2.1 | 1.4
  After First Vaccination, IM, Erythema-Mild: number analyzed (Participants) | 287 | 291 | 285
  After First Vaccination, IM, Erythema-Mild | 1.7 | 1.4 | 1.1
  After First Vaccination, IM, Erythema-Moderate: number analyzed (Participants) | 287 | 291 | 285
  After First Vaccination, IM, Erythema-Moderate | 0 | 0.3 | 0
  After First Vaccination, IM, Swelling-Any: number analyzed (Participants) | 285 | 291 | 285
  After First Vaccination, IM, Swelling-Any | 1.8 | 0.3 | 1.1
  After First Vaccination, IM, Swelling-Mild: number analyzed (Participants) | 285 | 291 | 285
  After First Vaccination, IM, Swelling-Mild | 1.4 | 0 | 0.7
  After First Vaccination, SC,Any Local AEs: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, SC,Any Local AEs | 15.6 | 47.3 | 47.0
  After First Vaccination SC, Pain-Any: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination SC, Pain-Any | 14.2 | 40.4 | 42.5
  After First Vaccination SC, Pain-Mild: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination SC, Pain-Mild | 12.5 | 35.6 | 36.1
  After First Vaccination, SC, Pain-Moderate: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, SC, Pain-Moderate | 1.7 | 4.8 | 6.3
  After First Vaccination, SC, Erythema-Any: number analyzed (Participants) | 286 | 291 | 285
  After First Vaccination, SC, Erythema-Any | 1.7 | 16.8 | 14.4
  After First Vaccination, SC, Erythema-Mild: number analyzed (Participants) | 286 | 291 | 285
  After First Vaccination, SC, Erythema-Mild | 1.0 | 15.8 | 12.3
  After First Vaccination, SC, Erythema-Moderate: number analyzed (Participants) | 286 | 291 | 285
  After First Vaccination, SC, Erythema-Moderate | 0 | 1.0 | 1.8
  After First Vaccination, SC, Swelling-Any: number analyzed (Participants) | 286 | 291 | 285
  After First Vaccination, SC, Swelling-Any | 1.0 | 2.7 | 2.8
  After First Vaccination, SC, Swelling-Mild: number analyzed (Participants) | 286 | 291 | 285
  After First Vaccination, SC, Swelling-Mild | 0.7 | 2.7 | 2.5
  After Second Vaccination, SC,Any Local AEs: number analyzed (Participants) | 255 | 264 | 251
  After Second Vaccination, SC,Any Local AEs | 11.0 | 37.9 | 41.0
  After Second Vaccination, SC,Pain-Any: number analyzed (Participants) | 255 | 262 | 251
  After Second Vaccination, SC,Pain-Any | 10.6 | 34.7 | 37.8
  After Second Vaccination, SC,Pain-Mild: number analyzed (Participants) | 255 | 262 | 251
  After Second Vaccination, SC,Pain-Mild | 10.2 | 30.9 | 33.9
  After Second Vaccination, SC,Pain-Moderate: number analyzed (Participants) | 255 | 262 | 251
  After Second Vaccination, SC,Pain-Moderate | 0.4 | 2.7 | 3.2
  After Second Vaccination, SC,Pain-Severe: number analyzed (Participants) | 255 | 262 | 251
  After Second Vaccination, SC,Pain-Severe | 0 | 1.1 | 0.8
  After Second Vaccination, SC,Erythema-Any: number analyzed (Participants) | 254 | 263 | 250
  After Second Vaccination, SC,Erythema-Any | 0.4 | 12.9 | 11.6
  After Second Vaccination, SC,Erythema-Mild: number analyzed (Participants) | 254 | 263 | 250
  After Second Vaccination, SC,Erythema-Mild | 0.4 | 12.2 | 10.0
  After Second Vaccination, SC,Erythema-Moderate: number analyzed (Participants) | 254 | 263 | 250
  After Second Vaccination, SC,Erythema-Moderate | 0 | 0.8 | 1.2
  After Second Vaccination, SC,Swelling-Any: number analyzed (Participants) | 254 | 263 | 249
  After Second Vaccination, SC,Swelling-Any | 0.8 | 4.6 | 4.8
  After Second Vaccination, SC,Swelling-Mild: number analyzed (Participants) | 254 | 263 | 249
  After Second Vaccination, SC,Swelling-Mild | 0.8 | 3.4 | 4.4
  After Second Vaccination, SC,Swelling-Moderate: number analyzed (Participants) | 254 | 263 | 249
  After Second Vaccination, SC,Swelling-Moderate | 0 | 0.8 | 0

6. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) by Severity After Each Vaccination
Description: Solicited systemic AEs include fever, headache, asthenia, malaise and myalgia that occurred within 14 days after each vaccination. Solicited systemic AEs (headache, asthenia, malaise and myalgia) was graded from 0 to 3 by severity; where 0=None, 1=Mild: No interference with daily activity, 2=Moderate: Interference with daily activity, 3=Severe: Prevents daily activity; A systemic AE of fever (defined as ≥38°C or ≥100.4°F) was derived from a daily temperature reading recorded within 14 days after vaccination. Fever was excluded from the overall count as no severity grading was applied for it. The percentages were rounded off to the first decimal place.
Time Frame: Within 14 days after each vaccination
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 299 | 300 | 298
percentage of participants
  After First Vaccination, Any Systemic AEs: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Any Systemic AEs | 47.4 | 44.2 | 49.5
  After First Vaccination, Headache-Any: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Headache-Any | 28.7 | 32.5 | 31.2
  After First Vaccination, Headache-Mild: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Headache-Mild | 19.0 | 22.3 | 20.7
  After First Vaccination, Headache-Moderate: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Headache-Moderate | 8.7 | 8.2 | 8.8
  After First Vaccination, Headache-Severe: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Headache-Severe | 1.0 | 2.1 | 1.8
  After First Vaccination, Asthenia-Any: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Asthenia-Any | 17.0 | 15.8 | 20.7
  After First Vaccination, Asthenia-Mild: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Asthenia-Mild | 12.8 | 9.2 | 16.1
  After First Vaccination, Asthenia-Moderate: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Asthenia-Moderate | 4.2 | 5.5 | 4.2
  After First Vaccination, Asthenia-Severe: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Asthenia-Severe | 0 | 1.0 | 0.4
  After First Vaccination, Malaise-Any: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Malaise-Any | 17.6 | 21.2 | 21.8
  After First Vaccination, Malaise-Mild: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Malaise-Mild | 11.4 | 13.7 | 14.0
  After First Vaccination, Malaise-Moderate: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Malaise-Moderate | 5.2 | 5.8 | 7.0
  After First Vaccination, Malaise-Severe: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Malaise-Severe | 1.0 | 1.7 | 0.7
  After First Vaccination, Myalgia-Any: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Myalgia-Any | 29.4 | 22.9 | 33.7
  After First Vaccination, Myalgia-Mild: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Myalgia-Mild | 23.9 | 16.4 | 27.7
  After First Vaccination, Myalgia-Moderate: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Myalgia-Moderate | 5.2 | 6.2 | 5.6
  After First Vaccination, Myalgia-Severe: number analyzed (Participants) | 289 | 292 | 285
  After First Vaccination, Myalgia-Severe | 0.3 | 0.3 | 0.4
  After First Vaccination, Fever-Any: number analyzed (Participants) | 289 | 292 | 284
  After First Vaccination, Fever-Any | 1.7 | 2.7 | 1.8
  After First Vaccination, Fever-38.0-<38.5: number analyzed (Participants) | 289 | 292 | 284
  After First Vaccination, Fever-38.0-<38.5 | 1.4 | 2.1 | 0.7
  After First Vaccination, Fever-38.5-<39.0: number analyzed (Participants) | 289 | 292 | 284
  After First Vaccination, Fever-38.5-<39.0 | 0.3 | 0.7 | 0.4
  After First Vaccination, Fever-39.0-<39.5: number analyzed (Participants) | 289 | 292 | 284
  After First Vaccination, Fever-39.0-<39.5 | 0 | 0 | 0.4
  After First Vaccination, Fever-≥41.0: number analyzed (Participants) | 289 | 292 | 284
  After First Vaccination, Fever-≥41.0 | 0 | 0 | 0.4
  After Second Vaccination, Any Systemic AEs: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Any Systemic AEs | 27.6 | 30.2 | 33.1
  After Second Vaccination, Headache-Any: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Headache-Any | 17.7 | 17.2 | 22.3
  After Second Vaccination, Headache-Mild: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Headache-Mild | 13.0 | 12.6 | 14.7
  After Second Vaccination, Headache-Moderate: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Headache-Moderate | 4.3 | 3.4 | 6.0
  After Second Vaccination, Headache-Severe: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Headache-Severe | 0.4 | 1.1 | 1.6
  After Second Vaccination, Asthenia-Any: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Asthenia-Any | 9.8 | 7.6 | 11.2
  After Second Vaccination, Asthenia-Mild: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Asthenia-Mild | 7.5 | 5.0 | 7.6
  After Second Vaccination, Asthenia-Moderate: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Asthenia-Moderate | 2.4 | 2.7 | 1.6
  After Second Vaccination, Asthenia-Severe: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Asthenia-Severe | 0 | 0 | 2.0
  After Second Vaccination, Malaise-Any: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Malaise-Any | 14.6 | 14.9 | 16.3
  After Second Vaccination, Malaise-Mild: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Malaise-Mild | 10.2 | 9.9 | 10.4
  After Second Vaccination, Malaise-Moderate: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Malaise-Moderate | 3.1 | 3.8 | 3.6
  After Second Vaccination, Malaise-Severe: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Malaise-Severe | 1.2 | 1.1 | 2.4
  After Second Vaccination, Myalgia-Any: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Myalgia-Any | 12.6 | 15.6 | 19.5
  After Second Vaccination, Myalgia-Mild: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Myalgia-Mild | 10.2 | 13.0 | 15.9
  After Second Vaccination, Myalgia-Moderate: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Myalgia-Moderate | 2.0 | 1.9 | 3.2
  After Second Vaccination, Myalgia-Severe: number analyzed (Participants) | 254 | 262 | 251
  After Second Vaccination, Myalgia-Severe | 0.4 | 0.8 | 0.4
  After Second Vaccination, Fever-Any: number analyzed (Participants) | 251 | 262 | 250
  After Second Vaccination, Fever-Any | 3.6 | 1.1 | 0.8
  After Second Vaccination, Fever-38.0-<38.5: number analyzed (Participants) | 251 | 262 | 250
  After Second Vaccination, Fever-38.0-<38.5 | 3.2 | 0.4 | 0.8
  After Second Vaccination, Fever-38.5-<39.0: number analyzed (Participants) | 251 | 262 | 250
  After Second Vaccination, Fever-38.5-<39.0 | 0 | 0.4 | 0
  After Second Vaccination, Fever-39.5-<40.0: number analyzed (Participants) | 251 | 262 | 250
  After Second Vaccination, Fever-39.5-<40.0 | 0.4 | 0.4 | 0

7. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs) After Each Vaccination
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration.
Time Frame: Up to 28 days (Day of Vaccination+27 Subsequent Days) after each vaccination
Population: Safety Set included all participants who received at least 1 dose of trial vaccine. Number analyzed is the number of participants with data available for the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 299 | 300 | 298
percentage of participants
  After First Vaccination | 14.7 | 17.0 | 18.8
  After Second Vaccination: number analyzed (Participants) | 270 | 271 | 257
  After Second Vaccination | 14.4 | 10.0 | 11.7

8. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: A SAE is defined as any untoward medical occurrence that: 1) results in death, 2) is life-threatening, 3) requires inpatient hospitalization or prolongation of existing hospitalization, 4) results in persistent or significant disability/incapacity, 5) leads to a congenital anomaly/birth defect in the offspring of the participant or 6) is an medically important event that satisfies any of the following: a) May require intervention to prevent items 1 through 5 above. b) May expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.
Time Frame: From the first vaccination on Day 1 until the end of the trial (Day 270)
Population: Safety Set included all participants who received at least 1 dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 299 | 300 | 298
percentage of participants | 0.7 | 2.7 | 2.3

9. Secondary Outcome: Percentage of Participants With Medically Attended AEs (MAAEs)
Description: MAAEs are defined as AEs leading to a medical visit to or by a healthcare professional, including visits to an emergency department, but not fulfilling seriousness criteria.
Time Frame: From the first vaccination on Day 1 until the end of the trial (Day 270)
Population: Safety Set included all participants who received at least 1 dose of trial vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
Number analyzed (Participants) | 299 | 300 | 298
percentage of participants | 23.1 | 21.0 | 20.1

ADVERSE EVENTS:
Time Frame: All-cause mortality and Serious adverse events: From the first vaccination on Day 1 until the end of the trial (Day 270); Other adverse events: Up to 28 days (Day of vaccination+27 subsequent days) after each vaccination.
Description: Safety Set included all participants who received at least 1 dose of trial vaccine.
Arm/Group | HAV Vaccine 1.0 ml + Placebo/ Placebo | TDV 0.5 ml + Placebo/ TDV 0.5 ml | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/300 | 0/298
Serious Adverse Events (participants affected / at risk) | 2/299 | 8/300 | 7/298
Other Adverse Events (participants affected / at risk) | 9/299 | 8/300 | 11/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HAV Vaccine 1.0 ml + Placebo/ Placebo (N=299) | TDV 0.5 ml + Placebo/ TDV 0.5 ml (N=300) | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml (N=298)
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HAV Vaccine 1.0 ml + Placebo/ Placebo (N=299) | TDV 0.5 ml + Placebo/ TDV 0.5 ml (N=300) | TDV 0.5 ml + HAV Vaccine 1.0 ml/ TDV 0.5 ml (N=298)
Nasopharyngitis (Infections and infestations) | 9 | 8 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT03525119/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT03525119/SAP_001.pdf